CLINICAL TRIAL: NCT05875805
Title: A Telehealth Advance Care Planning Intervention for Older Patients With Myeloid Malignancies: A Pilot Randomized Controlled Trial
Brief Title: A Telehealth Advance Care Planning Intervention
Acronym: SICP RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Kah Poh Loh, Associate Professor - Department of Medicine, Hematology/Oncology (SMD), University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UOCPC23038
Record Dates: First submitted 2023-05-16; First posted 2023-05-25 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Myeloid Malignancy; Acute Myeloid Leukemia; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasm; Myelofibrosis
Keywords: Older adults; Myeloid malignancies; Geriatric hematology; Serious illness conversations
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Primary Myelofibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telehealth Serious Illness Care Program (Experimental): The adapted telehealth Serious Illness Care Program is a multilevel intervention engaging the patient, caregiver, clinician, and system. It consists of tools, training, and system change. Tools include: 1) The Serious Illness Conversation Guide for clinicians; and 2) Education materials for patients on the importance of Serious Illness Conversations (Patient Preparation Pamphlet) and of the involvement of caregivers (Family Communication Guide).
  Interventions: Behavioral: Telehealth Serious Illness Care Program
- Control (Other): Education materials developed by the NCI on "Communication in Cancer Care (PDQ®) - Patient Version"
  Interventions: Other: Education Control

INTERVENTIONS:
Behavioral: Telehealth Serious Illness Care Program — The adapted telehealth Serious Illness Care Program is a multilevel intervention engaging the patient, caregiver, clinician, and system. It consists of tools, training, and system change. Tools include: 1) The Serious Illness Conversation Guide for clinicians; and 2) Education materials for patients on the importance of Serious Illness Conversations (Patient Preparation Pamphlet) and of the involvement of caregivers (Family Communication Guide).
  Arms: Telehealth Serious Illness Care Program
Other: Education Control — Education materials developed by the NCI on "Communication in Cancer Care (PDQ®) - Patient Version"
  Arms: Control

SUMMARY:
The objective of this project is to conduct a pilot randomized trial to assess the preliminary efficacy of a telehealth-delivered Serious Illness Care Program on healthcare communication, patient anxiety and distress, as well as completion of advance directives (specifically MOLST and healthcare proxy forms) for older patients with acute myeloid leukemia, myelodysplastic syndrome, and similar myeloid malignancies.

DETAILED DESCRIPTION:
The Serious Illness Care Program (SICP) is an evidence-based intervention to enhance serious illness conversations between physicians and patients with advanced cancer. It consists of the Serious Illness Conversation Guide as well as training and system-level support for clinicians to conduct serious illness conversations. The investigators have previously adapted the SICP to be delivered via telehealth for older adults with myeloid malignancies. In this study, they will conduct a pilot randomized trial to assess the preliminary efficacy of a telehealth-delivered Serious Illness Care Program compared to an education control.

ELIGIBILITY:
Inclusion and Exclusion Criteria for Patients

Inclusion criteria:

* Age ≥60 years
* A diagnosis of AML, MDS, and similar myeloid malignancies (including but not limited to MDS/MPN overlap syndrome, myelofibrosis)
* Being managed in the outpatient settings
* Able to provide informed consent
* English-speaking

Exclusion criteria:

- None

Inclusion and Exclusion Criteria for Caregivers

Inclusion criteria:

* Age ≥18 years
* Selected by patient when asked if there is a "family member, partner, friend, or caregiver with whom you discuss or who can be helpful in health-related matters"
* Able to provide informed consent
* English-speaking

Exclusion criteria:

- None

Inclusion and Exclusion Criteria for Oncology Providers

Inclusion criteria:

- Oncologists and/or APPs who will be conducting the telehealth-delivered ACP visit

Exclusion criteria:

- None

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Estimated)
Dates: Start 2024-05-20 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Healthcare Communication: Health Care Climate Questionnaire | Month 2
  5-item questionnaire assessing patients' and caregivers' satisfaction with patient-clinician communication, range 0-20; higher score is better

SECONDARY OUTCOMES:
Distress: Distress Thermometer | Month 2
  1-item question for distress, range 0-10; higher scores indicate greater distress
Anxiety Symptoms: Generalized Anxiety Disorder-7 (GAD-7) | Month 2
  7-item screening tool for anxiety symptoms, total range 0-21); higher scores indicate greater anxiety symptoms
Completion of advance directives | Throughout the study, up to 2 years
  Percentage of patients who complete advance directives which include the Medical or Physician Orders for Life-Sustaining Treatment (MOST/POLST) forms, living will, durable power of attorney for healthcare, and healthcare proxy forms, as well as date of completion

CONTACTS AND LOCATIONS:
Overall Officials: Kah Poh Loh, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared with other investigators if requested. Published papers will be made available in portable document format.
Supporting Information: Study Protocol
Time Frame: The data will be available for 7 years after study completion

REFERENCES:
- [Background] LoCastro M, Sanapala C, Mendler JH, Norton S, Bernacki R, Carroll T, Klepin HD, Watson E, Liesveld J, Huselton E, O'Dwyer K, Baran A, Flannery M, Kluger B, Loh KP. Adaptation of Serious Illness Care Program to be delivered via telehealth for older patients with hematologic malignancy. Blood Adv. 2023 May 9;7(9):1871-1884. doi: 10.1182/bloodadvances.2022008996. PMID 36521100
- [Background] LoCastro M, Sanapala C, Mendler JH, Norton S, Bernacki R, Carroll T, Klepin H, Watson E, Liesveld J, Huselton E, O'Dwyer K, Baran A, Flannery M, Kluger BM, Loh KP. Advance care planning in older patients with acute myeloid leukemia and myelodysplastic syndromes. J Geriatr Oncol. 2023 Jan;14(1):101374. doi: 10.1016/j.jgo.2022.09.003. Epub 2022 Sep 10. PMID 36100548